CLINICAL TRIAL: NCT01849887
Title: Safety of Escalating Doses of Intravenous Bone Marrow-Derived Mesenchymal Stem Cells in Patients With a New Ischemic Stroke
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was never started
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR3-07521
Record Dates: First submitted 2013-05-06; First posted 2013-05-09 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mesenchymal stem cells (Active Comparator): bone marrow-derived mesenchymal stem cells
  Interventions: Biological: bone marrow-derived mesenchymal stem cells
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: bone marrow-derived mesenchymal stem cells — bone marrow-derived mesenchymal stem cells
  Arms: mesenchymal stem cells
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Stroke is a major cause of adult disability. Currently approved reperfusion therapies are provided to only a small percentage of patients in the U.S. New therapies are needed that improve outcome and that can be accessed by a majority of patients. Animal studies suggest that bone marrow-derived mesenchymal stem cells, administered intravenously days after a stroke, safely improve long-term behavioral outcome. A large human experience suggests the safety of allogeneic bone marrow-derived mesenchymal stem cells. The current study aims to assess the safety of this therapy in patients with recent ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ischemic stroke in the middle cerebral artery territory, with onset 24-72 hours prior to the time that the therapy transfusion is initiated, radiologically confirmed, and with either diameter >15 mm or volume > 4cc.
* 2. The index stroke has clinical deficits that are moderate-severe (NIHSS score 7-20), did not require hemicraniectomy or invasive intracranial pressure monitoring, and was not associated with a concomitant STelevation myocardial infarction.
* 3. Age 18-80 years, inclusive
* 4. Reasonable likelihood of receiving standard post-stroke medical care, as well as standard physical, occupational, and speech therapy.

Exclusion Criteria:

* 1. No substantial pre-stroke disability (pre-stroke modified Rankin Scale score 0-2).
* 2. Females of child-bearing potential will be excluded unless (1) a negative urine pregnancy test is obtained and (2) the patient has been effectively using contraceptive method with known failure rate <1 % for at least 90 days.
* 3. Lactating mothers
* 4. If thrombolytic therapy has been administered, at least 24 hours have passed between completing thrombolytic dosing and initiating the current study's transfusion.
* 5. Known allergy to penicillin or to fetal bovine serum
* 6. Active co-existent major neurological or psychiatric disease that could significantly interfere with patient compliance or study assessments, including drug or alcohol abuse.
* 7. Any diagnosis that makes survival to 1-year post-stroke unlikely.
* 8. Participation in any other experimental therapeutic clinical trial concurrently or in the prior three months.
* 9. Contraindication to undergoing MRI scanning.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 1 month after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Steve Cramer, MD, Principal Investigator — Univ Calif Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States